CLINICAL TRIAL: NCT03157713
Title: Financial Incentive Strategies for Weight Loss in Obese Patients Living in Socioeconomically Disadvantaged Neighborhoods
Brief Title: Financial Incentives for Weight Reduction Study
Acronym: FIReWoRk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Soma Wali, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01MD011544-03 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Obese
Keywords: Obesity; Weight-loss; Financial Incentives; Behavioral Economics
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Goal-Directed (Experimental): Patients will receive enhanced usual care and also be informed that they will receive goal-directed financial incentives.
  Interventions: Behavioral: Goal-Directed Financial Incentives; Behavioral: Enhanced Usual Care
- Outcome-Based (Experimental): Patients will receive enhanced usual care and be informed that they will receive outcome-based financial incentives for significant weight losses.
  Interventions: Behavioral: Enhanced Usual Care; Behavioral: Outcome-based Financial Incentives
- Control-Enhanced Usual Care (Other): Patients will only receive enhanced usual care.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Goal-Directed Financial Incentives — Patients will receive financial incentives for using a food diary, verified by entries in in the BookFactory Food Diary or another food diary, including internet/app-based diaries ($30 monthly); achieving 75 minutes of physical activity per week in first three months, as verified by a wearable fitness tracker ($20 monthly); achieving 150 minutes of physical activity per week in last three months, as verified by a wearable fitness tracker ($20 monthly); enrollment in a clinic-based or commercial weight loss program ($150 one time); and active participation in clinic-based or commercial weight loss program, as verified by the program ($60 monthly).
  Arms: Goal-Directed
Behavioral: Enhanced Usual Care — Patients will receive a food diary (BookFactory Food Diary), wearable fitness tracker (Fitbit), exercise and nutrition education materials (American Heart Association's Walking For Better Health and How to Eat Healthy), and referral information for intensive weight loss programs. This information will comprise these commercial and hospital-based weight loss programs that are evidence-based: Weight Watchers and Jenny Craig; the Veterans Administration's MOVE! and TeleMOVE! programs; Bellevue Hospital's Medical Weight Management Clinic and Intensive Nutritional Treatment programs; and New York University Langone Medical Center's Weight Management Program. We will also provide brief instructions on how to use the food diary and Fitbit Charge HR.
Behavioral: Outcome-based Financial Incentives — Patients will receive financial incentives for clinically significant weight loss, as confirmed at monthly weigh-ins. At 30 days, they will receive $50 if they lose ≥1.5% to <2.5% of baseline weight or $100 if they lose ≥2.5% of baseline weight. At 2 months and 3 months, they will receive $50 if they lose ≥2.5% to <5% of baseline weight or $100 if they lose ≥5% of baseline weight. At 4, 5, and 6 months, they will receive $100 if they lose ≥2.5% to <5% of baseline weight or $150 if they lose ≥5% of baseline weight. To employ the behavioral economic concept of regret aversion, patients will be given feedback at each assessment point about incentives they would have received had they achieved a loss of at least 2.5% of baseline weight.
  Arms: Outcome-Based

SUMMARY:
Financial incentives for motivating changes in health behavior, particularly for weight loss in obese individuals, are increasingly being tested by health insurers, employers, and government agencies. However, a key unanswered question regarding weight loss is how to structure these incentive programs to maximize their effectiveness, acceptability to patients, and economic sustainability. Focusing on obese patients living in neighborhoods with a high concentration of low socioeconomic status households, the investigators will compare the impact of financial incentives for weight loss on sustained weight loss, use of evidenced-based therapy, and quality of life, and they will determine their short-term and long-term return on investment.

DETAILED DESCRIPTION:
Financial incentives for motivating changes in health behavior, for weight loss in obese individuals, are increasingly being tested by health insurers, employers, and government agencies. However, a key unanswered question regarding weight loss is how to structure these incentive programs to maximize their (1) effectiveness, underscored by the fact that most programs have not resulted in significant long-term weight loss; and (2) economic sustainability, as defined by their return on investment-a major factor in public and private decision-making.

Obese patients represent an important population to target for effective weight loss interventions because they suffer from a high prevalence of serious obesity-related illnesses-including diabetes, hypertension, dyslipidemia, heart disease, stroke, sleep apnea, and cancer-disproportionately have a low socioeconomic status, and impose $147 billion in costs on the healthcare system annually. While prior studies testing financial incentives in this population have had variable short-term success and few have yielded long-term weight loss, a fundamental question remains unanswered and may partially explain variability in weight loss outcomes: specifically, it is unknown whether goal-directed incentives (incentives for achieving evidence-based, intermediate goals that increase weight loss but are underutilized, like dietary counseling, physical activity, behavioral self-monitoring, and intensive weight management programs) or outcome-based incentives (like incentives for successfully losing weight) are more effective for promoting weight loss. Prior studies of weight loss incentives have largely emphasized only the latter.

The investigators propose a three-arm randomized controlled trial that will address this important knowledge gap among obese patients living in socioeconomically disadvantaged neighborhoods, with implications for other serious chronic health conditions. Comparing goal-directed incentives to outcome-based incentives and usual care, the investigators will assess their impact on weight loss (≥5% of baseline weight), use of evidenced-based therapy, and quality of life, and evaluate their short-term and long-term return on investment.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking patients
* Under the care of a primary care physician at Manhattan VA, Bellevue, NYU Langone Medical Center, or Olive View-UCLA Medical Center
* With obesity, based on BMI of 30 to 40 kg/m2 during a prior visit in the past 6 months
* Who are between the age of 18 and 70 years
* Who have an active U.S. phone number and address

Exclusion Criteria:

* have had weight loss ≥4.5 kg
* participated in an intensive weight loss program in the past 6 mo.
* abuse alcohol/other substances
* have active psychosis/other cognitive issues
* have history of myocardial infarction/stroke in the past 6 mo. or metastatic cancer
* New York Heart Association Class III/IV heart failure
* Chronic Kidney Disease stage IV/V
* pregnant or breastfeeding or plan to become pregnant within subsequent 12 mo.
* have history of an eating disorder/unsafe weight-loss behaviors
* are unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve 5% reduction from Baseline Weight at 6 months | Baseline and 6 months
  We will obtain weight measurements by weighing before eating without shoes or heavy garments using a digital scale that will be calibrated monthly.

SECONDARY OUTCOMES:
Change in quality of life measured by 12-Item Short Form Survey (Version 2). | Baseline and 6 months
  Assessed using SF-12v2 survey.
Change in Quality of Life Measured by EQ5-5D-5L | Baseline and 6 months
  Assessed using EQ-5D-5L questionnaire.
Changes in Waist Circumference | Baseline, 6 Months, 9 Months and 12 Months
  Measured using a standard tape measure
Changes in Blood Pressure | Baseline, 6 Months, 9 Months and 12 Months
  Assessed using an automated sphygmomanometer
Use of evidenced-based weight loss programs assessed by documentation of enrollment. | 6 months
  Patients will have the option to either (1) provide consent for the investigators to contact and confirm enrollment and participation in evidence-based, commercial weight loss programs, or (2) procure documentation to confirm enrollment and participation.
Short term return on investment of using financial incentives to promote weight loss | 9 months
  Cost analysis involving hospital utilization data, electronic health records, patient reported healthcare utilization, and micro-simulation modeling.
Long term return on investment of using financial incentives to promote weight loss | 12 months
  Cost analysis involving hospital utilization data, electronic health records, patient reported healthcare utilization, and micro-simulation modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Ladapo, MD./PhD., Principal Investigator — University of California, Los Angeles; Melanie Jay, MD., Principal Investigator — New York University
Locations (2):
- United States (2):
  - Olive View-UCLA Medical Center, Sylmar, California
  - NYU Lutheran Medical Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gudzune KA, Doshi RS, Mehta AK, Chaudhry ZW, Jacobs DK, Vakil RM, Lee CJ, Bleich SN, Clark JM. Efficacy of commercial weight-loss programs: an updated systematic review. Ann Intern Med. 2015 Apr 7;162(7):501-12. doi: 10.7326/M14-2238. PMID 25844997
- [Background] Eckel RH, Jakicic JM, Ard JD, de Jesus JM, Houston Miller N, Hubbard VS, Lee IM, Lichtenstein AH, Loria CM, Millen BE, Nonas CA, Sacks FM, Smith SC Jr, Svetkey LP, Wadden TA, Yanovski SZ, Kendall KA, Morgan LC, Trisolini MG, Velasco G, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S76-99. doi: 10.1161/01.cir.0000437740.48606.d1. Epub 2013 Nov 12. No abstract available. PMID 24222015
- [Background] Boutelle KN, Kirschenbaum DS. Further support for consistent self-monitoring as a vital component of successful weight control. Obes Res. 1998 May;6(3):219-24. doi: 10.1002/j.1550-8528.1998.tb00340.x. PMID 9618126
- [Background] Brazier JE, Roberts J. The estimation of a preference-based measure of health from the SF-12. Med Care. 2004 Sep;42(9):851-9. doi: 10.1097/01.mlr.0000135827.18610.0d. PMID 15319610
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Murphy SL. Review of physical activity measurement using accelerometers in older adults: considerations for research design and conduct. Prev Med. 2009 Feb;48(2):108-14. doi: 10.1016/j.ypmed.2008.12.001. Epub 2008 Dec 10. PMID 19111780
- [Background] Strickland S. Does it work to pay people to live healthier lives? BMJ. 2014 Apr 2;348:g2458. doi: 10.1136/bmj.g2458. No abstract available. PMID 24696175
- [Background] Towers Watson National Business Group on Health. Full Report: Towers Watson/NBGH 2013/2014 Employer Survey on Purchasing Value in Health Care. 2014; http://www.towerswatson.com/en-US/Insights/IC-Types/Survey-Research-Results/2014/05/full-report-towers-watson-nbgh-2013-2014-employer-survey-on-purchasing-value-in-health-care. Accessed August 4, 2015.
- [Background] Leatherman S, Berwick D, Iles D, Lewin LS, Davidoff F, Nolan T, Bisognano M. The business case for quality: case studies and an analysis. Health Aff (Millwood). 2003 Mar-Apr;22(2):17-30. doi: 10.1377/hlthaff.22.2.17. PMID 12674405
- [Background] Nguyen NT, Magno CP, Lane KT, Hinojosa MW, Lane JS. Association of hypertension, diabetes, dyslipidemia, and metabolic syndrome with obesity: findings from the National Health and Nutrition Examination Survey, 1999 to 2004. J Am Coll Surg. 2008 Dec;207(6):928-34. doi: 10.1016/j.jamcollsurg.2008.08.022. Epub 2008 Oct 10. PMID 19183541
- [Background] Haslam DW, James WP. Obesity. Lancet. 2005 Oct 1;366(9492):1197-209. doi: 10.1016/S0140-6736(05)67483-1. PMID 16198769
- [Background] Drewnowski A, Rehm CD, Solet D. Disparities in obesity rates: analysis by ZIP code area. Soc Sci Med. 2007 Dec;65(12):2458-63. doi: 10.1016/j.socscimed.2007.07.001. Epub 2007 Aug 29. PMID 17761378
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] John LK, Loewenstein G, Troxel AB, Norton L, Fassbender JE, Volpp KG. Financial incentives for extended weight loss: a randomized, controlled trial. J Gen Intern Med. 2011 Jun;26(6):621-6. doi: 10.1007/s11606-010-1628-y. Epub 2011 Jan 20. PMID 21249462
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Jolly K, Lewis A, Beach J, Denley J, Adab P, Deeks JJ, Daley A, Aveyard P. Comparison of range of commercial or primary care led weight reduction programmes with minimal intervention control for weight loss in obesity: lighten Up randomised controlled trial. BMJ. 2011 Nov 3;343:d6500. doi: 10.1136/bmj.d6500. PMID 22053315
- [Background] Kullgren JT, Troxel AB, Loewenstein G, Asch DA, Norton LA, Wesby L, Tao Y, Zhu J, Volpp KG. Individual- versus group-based financial incentives for weight loss: a randomized, controlled trial. Ann Intern Med. 2013 Apr 2;158(7):505-14. doi: 10.7326/0003-4819-158-7-201304020-00002. PMID 23546562
- [Background] Patel MS, Asch DA, Troxel AB, Fletcher M, Osman-Koss R, Brady J, Wesby L, Hilbert V, Zhu J, Wang W, Volpp KG. Premium-Based Financial Incentives Did Not Promote Workplace Weight Loss In A 2013-15 Study. Health Aff (Millwood). 2016 Jan;35(1):71-9. doi: 10.1377/hlthaff.2015.0945. PMID 26733703
- [Background] Finkelstein EA, Linnan LA, Tate DF, Birken BE. A pilot study testing the effect of different levels of financial incentives on weight loss among overweight employees. J Occup Environ Med. 2007 Sep;49(9):981-9. doi: 10.1097/JOM.0b013e31813c6dcb. PMID 17848854
- [Background] Garcia DO, Jakicic JM, Davis KK, Gibbs BB, Burke LE, Rickman AD. A Pilot Feasibility Study of a Campaign Intervention for Weight Loss among Overweight and Obese Adults. 2014.
- [Background] Leahey T, Rosen J. DietBet: A Web-Based Program that Uses Social Gaming and Financial Incentives to Promote Weight Loss. JMIR Serious Games. 2014 Feb 7;2(1):e2. doi: 10.2196/games.2987. PMID 25658966
- [Background] Leahey TM, Subak LL, Fava J, Schembri M, Thomas G, Xu X, Krupel K, Kent K, Boguszewski K, Kumar R, Weinberg B, Wing R. Benefits of adding small financial incentives or optional group meetings to a web-based statewide obesity initiative. Obesity (Silver Spring). 2015 Jan;23(1):70-6. doi: 10.1002/oby.20937. Epub 2014 Nov 11. PMID 25384463
- [Background] Moller AC, McFadden HG, Hedeker D, Spring B. Financial motivation undermines maintenance in an intensive diet and activity intervention. J Obes. 2012;2012:740519. doi: 10.1155/2012/740519. Epub 2012 Apr 2. PMID 22548152
- [Background] Spring B, Schneider K, McFadden HG, Vaughn J, Kozak AT, Smith M, Moller AC, Epstein LH, Demott A, Hedeker D, Siddique J, Lloyd-Jones DM. Multiple behavior changes in diet and activity: a randomized controlled trial using mobile technology. Arch Intern Med. 2012 May 28;172(10):789-96. doi: 10.1001/archinternmed.2012.1044. PMID 22636824
- [Derived] Ladapo JA, Orstad SL, Wali S, Wylie-Rosett J, Tseng CH, Chung UYR, Cuevas MA, Hernandez C, Parraga S, Ponce R, Sweat V, Wittleder S, Wallach AB, Shu SB, Goldstein NJ, Jay M. Effectiveness of Goal-Directed and Outcome-Based Financial Incentives for Weight Loss in Primary Care Patients With Obesity Living in Socioeconomically Disadvantaged Neighborhoods: A Randomized Clinical Trial. JAMA Intern Med. 2023 Jan 1;183(1):61-69. doi: 10.1001/jamainternmed.2022.5618. PMID 36469353
- [Derived] Jay M, Orstad SL, Wali S, Wylie-Rosett J, Tseng CH, Sweat V, Wittleder S, Shu SB, Goldstein NJ, Ladapo JA. Goal-directed versus outcome-based financial incentives for weight loss among low-income patients with obesity: rationale and design of the Financial Incentives foR Weight Reduction (FIReWoRk) randomised controlled trial. BMJ Open. 2019 Apr 8;9(4):e025278. doi: 10.1136/bmjopen-2018-025278. PMID 30962231